CLINICAL TRIAL: NCT00415077
Title: A Prospective Comparison of Photorefractive Keratectomy (PRK), PRK With Mitomycin-C and Laser Subepithelial Keratomileusis (LASEK) in the Treatment of Moderate and High Myopia
Brief Title: A Comparison of Photorefractive Keratectomy (PRK), PRK With Mitomycin-C and Laser Subepithelial Keratomileusis (LASEK) in the Treatment of Moderate and High Myopia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in excimer laser systems prior to completion of study
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency); C.R.Darnall Army Medical Center (U.S. Federal Agency); Blanchfield Army Community Hospital (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAMC WU# 04-23009
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: MODERATE AND HIGH MYOPIA
MeSH Terms: interventions — Keratectomy, Subepithelial, Laser-Assisted

ARMS (3):
- 2 (Active Comparator): LASEK- laser-assisted subepithelial keratectomy
  Interventions: Procedure: MMC PRK
- 3 (Active Comparator): Mitomycin C PRK
  Interventions: Procedure: LASEK
- 1 (Active Comparator): PRK- Photorefractive keratectomy
  Interventions: Procedure: PRK

INTERVENTIONS:
Procedure: PRK — PRK
  Arms: 1
Procedure: MMC PRK — mitomycin C PRK
  Arms: 2
Procedure: LASEK — LASEK
  Arms: 3

SUMMARY:
The purpose of this study is to assess whether there is a significant difference in visual outcomes or corneal haze after surface ablation for moderate and high myopia in active duty service members treated with PRK, Mitomycin-C (MMC) PRK and LASEK.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Normal, healthy, active duty adults age 21 years or older. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
3. Manifest refractive spherical equivalent of greater than -4.00 diopters (D) up to -10.00 D.
4. Best spectacle corrected visual acuity of 20/20 or better in both eyes.
5. Demonstrated refractive stability, confirmed by clinical records. Neither the spherical nor the cylindrical portion of the refraction may have changed more than 0.50D during the 12-month period immediately preceding the baseline examination, as confirmed by clinical records.
6. Both eyes must fall in the same refraction group and there must be less than 1 D difference between eyes.
7. Soft contact lens users must have removed their lenses at least 2 weeks before baseline measurements. Hard contact lens users (PMMA or rigid gas permeable lenses) must have removed their lenses at least 4 weeks prior to baseline measurements and have 2 central keratometry readings and 2 manifest refractions taken at least 1 week apart that do not differ by more than 0.50 D in either meridian.
8. Access to transportation to meet the follow-up requirements.
9. Available for evaluation during the 1-year follow-up period.
10. Consent of the subject's command to participate in the study.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding or intend to become pregnant during the study. Women of childbearing age will take a urine pregnancy test before starting this study.
2. Residual, recurrent or active ocular diseases or corneal abnormalities in either eye such as keratoconus, iritis, uveitis, keratoconjunctivitis sicca, vernal conjunctivitis, lagophthalmos, corneal scarring, glaucoma, previous steroid responder, occludable chamber angles, visually significant cataracts.
3. Medical condition(s), which, in the judgment of the investigator, may impair healing, including but not limited to: collagen vascular disease, autoimmune disease, immunodeficiency diseases, and ocular herpes zoster or simplex.
4. Concurrent topical or systemic medications that may impair healing, including corticosteroids, antimetabolites, isotretinoin (Accutane), amiodarone hydrochloride (Cordarone) and/or sumatripin (Imitrex).
5. Any physical or mental impairment that would preclude participation in any of the examinations.
6. Prior refractive or ocular surgery.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2004-06

PRIMARY OUTCOMES:
Efficacy in terms of uncorrected visual acuity and post operative refraction. Safety in terms of maintenance of best spectacle corrected acuity within 2 lines of preoperative levels. | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: KRAIG S BOWER, MD, Principal Investigator — DIRECTOR, CENTER FOR REFRACTIVE SURGERY WALTER REED ARMY MEDICAL CENTER
Locations (1):
- Walter Reed Army Medical Center, Center For Refractive Surgery, Washington D.C., District of Columbia, United States